CLINICAL TRIAL: NCT04181489
Title: A Phase II, Prospective, Multi-center Study of Sintilimab in Combination With R-CHOP in Patients With Treatment-naive EBV-positive DLBCL, NOS
Brief Title: Sintilimab in Combination With R-CHOP in Patients With Treatment-naive EBV-positive DLBCL, NOS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-SR-271
Record Dates: First submitted 2019-11-24; First posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: EBV-Positive DLBCL, Nos
Keywords: Sintilimab; R-CHOP; EBV-Positive DLBCL, nos; treatment-naive
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic | interventions — sintilimab; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab + R-CHOP (Experimental)
  Interventions: Drug: Sintilimab; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg d0
Drug: Rituximab — Rituximab 375 mg/m2 d0
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m2 d1
Drug: Doxorubicin — Doxorubicin 50 mg/m2 d1
Drug: Vincristine — Vincristine 1.4mg/m2 (maximum 2mg) d1
Drug: Prednisolone — Prednisolone 60mg/m2 d1-5

SUMMARY:
The prognosis of EBV+ DLBCL is dismal. Previous study showed that high level of PD-L1 expression in EBV+ DLBCL. The investigators therefore design this phase II study to investigate the safety and efficacy of sintilimab (an anti-PD-1 antibody) in combination with R-CHOP in patients with treatment-naive EBV+ DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed EBV-positive diffuse large B cell lymphoma, NOS, according to WHO 2016 criteria.

2. Understand and voluntarily sign an informed consent form, able to adhere to the study visit schedule and other protocol requirements.

3. Undergo whole-body PET/CT scan 28 days before enrolment and have a measurable or evaluable disease (nodal lesion: diameter ≥ 1.5cm; extranodal lesion≥1.0cm）according to Lugano 2014 criteria； 4. ECOG PS 0- 2; 5. Adequate organ function, defined as:

1. Blood routine test: neutrophil count ≥ 1.0×10⁹/L, platelet count ≥ 50×10⁹/L, hemoglobulin ≥8.0g/dL, without G-CSF usage or blood infusion within 7 days before examination.
2. Hepatic function: total bilirubin less than 1.5-fold of upper normal level; ALT and AST less than 2-fold of upper normal level.
3. Renal function: Serum creatine less than 1.5-fold of upper normal level or Ccr ≥ 50 mL/min.
4. Cardiac function: New York Heart Association class II or below (EF≥ 50% according to TDE)
5. Coagulative function: INR less than 1.5-fold of upper normal level, APTT less than 10s above upper normal level and PT less than 3s above upper normal level;
6. Thyroid function: normal baseline TSH level, or abnormal baseline TSH but normal T3/T4 level without symptoms; 6. Expected survival ≥ 3 months; 7. Age 18~70 years; 8. Female subjects in childbearing age, their serum or urine pregnancy test must be negative. All patients must agree to take effective contraceptive measures during treatment and 90 days after treatment.

Exclusion Criteria:

1. CNS or meningeal involvement;
2. Patients with secondary tumour, excluding cured (5 years without relapse) in situ Non-melanoma skin cancer. superficial bladder cancer, in situ cervical cancer, Gastrointestinal intramucous carcinoma and breast cancer;
3. Known sensitivity or allergy to investigational product;
4. Previous exposure to anti PD-1 antibody, anti PD-L1 antibody, anti PD-L2 antibody, anti CTLA-4 antibody, CAR-T therapy or any T cell co-stimulating antibody or checkpoint inhibitor;
5. Previous allogeneic organ transplantation or allogeneic stem cell transplantation;
6. Intention to use any other anti-tumour therapy during treatment;
7. Use of systemic anti-tumour treatment within 3 months before first dose of study regimen;
8. Active and severe infectious diseases requiring systemic treatment;
9. Active (known or suspected) autoimmune disease or history of autoimmune disease within 2 years before treatment (excluding patients with leukoderma, psoriasis, lipsotrichia or Grave's disease who do not require systemic treatment within 2 years, patients with hypothyrea only requiring thyroxine as treatment, and patients with type I diabetes but only requiring insulin treatment)
10. Usage of immune inhibitory drugs 4 weeks before the first dose of study regimen, excluding local usage of glucocorticoid and systemic usage of less than 10mg/d Prednisone or equivalent glucocorticoid.
11. Active hepatitis B or hepatitis C virus infection, as well as acquired, congenital immune deficiency diseases, including but not limited to HIV-infected persons;
12. Previous history of Idiopathic pulmonary fibrosis or Idiopathic pneumonia;
13. Active tuberculosis;
14. Presence of ≥ Grade 3 immune therapy related toxicity;
15. History of mental disorder including epilepsia and dementia;
16. Any anti-infectious vital vaccine usage 4 weeks before the first dose or during treatment;
17. Any potential drug abuse, medical, psychological or social conditions which may disturb this investigation and assessment;
18. Women who are pregnant or lactating.
19. Usage of other experimental drugs within 1 month before treatment;
20. In any conditions which investigator considered ineligible for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Progressive free survival | 2 years
  from date of inclusion to date of progression, relapse, or death from any cause

SECONDARY OUTCOMES:
Overall response rate | 6 months
  overall response rate after treated by Sintilimab and R-CHOP
Overall survival | 2 years
  from the date of inclusion to date of death, irrespective of cause
Incidence of treatment related adverse events as assessed by NCI-CTCAE 5.0 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, M.D., Ph.D., Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital)
Locations (11):
- China (11):
  - ChangZhou First People's Hospital, Changzhou, Jiangsu
  - ChangZhou No.2 People's Hospital, Changzhou, Jiangsu
  - HuaiAn First People's Hospital, HuaiAn, Jiangsu
  - Drum tower hospital, Nanjing, Jiangsu
  - The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital), Nanjing, Jiangsu
  - The First Affiliated Hospital Of Nantong University, Nantong, Jiangsu
  - The Second Affiliated Hospital Of Suzhou University, Suzhou, Jiangsu
  - WuXi People's Hospital, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Yancheng First People's Hospital, Yancheng, Jiangsu
  - ZhenJiang First People's Hospital, Zhenjiang, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Swerdlow SH, Campo E, Pileri SA, Harris NL, Stein H, Siebert R, Advani R, Ghielmini M, Salles GA, Zelenetz AD, Jaffe ES. The 2016 revision of the World Health Organization classification of lymphoid neoplasms. Blood. 2016 May 19;127(20):2375-90. doi: 10.1182/blood-2016-01-643569. Epub 2016 Mar 15. PMID 26980727
- [Background] Coiffier B, Thieblemont C, Van Den Neste E, Lepeu G, Plantier I, Castaigne S, Lefort S, Marit G, Macro M, Sebban C, Belhadj K, Bordessoule D, Ferme C, Tilly H. Long-term outcome of patients in the LNH-98.5 trial, the first randomized study comparing rituximab-CHOP to standard CHOP chemotherapy in DLBCL patients: a study by the Groupe d'Etudes des Lymphomes de l'Adulte. Blood. 2010 Sep 23;116(12):2040-5. doi: 10.1182/blood-2010-03-276246. Epub 2010 Jun 14. PMID 20548096
- [Background] Ahn JS, Yang DH, Duk Choi Y, Jung SH, Yhim HY, Kwak JY, Sung Park H, Shin MG, Kim YK, Kim HJ, Lee JJ. Clinical outcome of elderly patients with Epstein-Barr virus positive diffuse large B-cell lymphoma treated with a combination of rituximab and CHOP chemotherapy. Am J Hematol. 2013 Sep;88(9):774-9. doi: 10.1002/ajh.23507. Epub 2013 Jul 23. PMID 23760676
- [Background] Sato A, Nakamura N, Kojima M, Ohmachi K, Carreras J, Kikuti YY, Numata H, Ohgiya D, Tazume K, Amaki J, Moriuchi M, Miyamoto M, Aoyama Y, Kawai H, Ichiki A, Hara R, Kawada H, Ogawa Y, Ando K. Clinical outcome of Epstein-Barr virus-positive diffuse large B-cell lymphoma of the elderly in the rituximab era. Cancer Sci. 2014 Sep;105(9):1170-5. doi: 10.1111/cas.12467. Epub 2014 Sep 8. PMID 24974976
- [Background] Hong JY, Yoon DH, Suh C, Huh J, Do IG, Sohn I, Jo J, Jung SH, Hong ME, Yoon H, Ko YH, Kim SJ, Kim WS. EBV-positive diffuse large B-cell lymphoma in young adults: is this a distinct disease entity? Ann Oncol. 2015 Mar;26(3):548-55. doi: 10.1093/annonc/mdu556. Epub 2014 Dec 4. PMID 25475080
- [Background] Lu TX, Liang JH, Miao Y, Fan L, Wang L, Qu XY, Cao L, Gong QX, Wang Z, Zhang ZH, Xu W, Li JY. Epstein-Barr virus positive diffuse large B-cell lymphoma predict poor outcome, regardless of the age. Sci Rep. 2015 Jul 23;5:12168. doi: 10.1038/srep12168. PMID 26202875
- [Background] Xu-Monette ZY, Zhou J, Young KH. PD-1 expression and clinical PD-1 blockade in B-cell lymphomas. Blood. 2018 Jan 4;131(1):68-83. doi: 10.1182/blood-2017-07-740993. Epub 2017 Nov 8. PMID 29118007